CLINICAL TRIAL: NCT03151499
Title: Effect of Rifampicin on the Pharmacokinetics of BI 409306 Following Oral Administration in Healthy Male Subjects (an Open-label, Two-period, Fixed Sequence Trial)
Brief Title: Drug-drug Interaction Trial Between Rifampicin and BI 409306 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1289-0044; 2016-004828-37 (EudraCT Number)
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 409306 (R), then BI 409306 after pretreatment with rifampicin (T) (Experimental): Subjects were administered during Period 1 on Day 1/Visit 2 a single dose of 50 milligrams (mg) of BI 409306 film-coated tablet orally with 240 millilitre (mL) of water (reference treatment, R).
  On Days -7 to -1 /Visit 3 of Period 2 participants were administered rifampicin 600 mg Eremfat® film-coated tablet orally with 240 mL of water once per day during the evenings. Afterwards on Day 1/Visit 3, participants were administered a single dose of 50 mg BI 409306 orally approximately 14 hours after the last rifampicin dose (test treatment, T).
  Due to the short half-life of BI 409306, trial period 2 directly followed trial period 1 without a wash-out period.
  Interventions: Drug: BI 409306; Drug: Rifampicin

INTERVENTIONS:
Drug: BI 409306 — Reference and Test Treatment
Drug: Rifampicin — Test Treatment

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of BI 409306 tablets with prior 7-day intake of rifampicin tablets (Test, T) compared to BI 409306 tablets without prior administration of rifampicin (Reference, R) following oral administration in healthy male subjects.

The secondary objective is the evaluation and comparison of several pharmacokinetic parameters between the treatments. The secondary objectives will be assessed by descriptive statistics.

ELIGIBILITY:
Inclusion criteria

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria

* Any finding in the medical examination (including (Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Current smoker or ex-smoker who quit smoking less than 30 days prior to screening.
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* History of relevant liver diseases such as disturbance of liver function, jaundice, drug induced liver injury, Dubin-Johnson syndrome, Rotor syndrome, or liver tumours
* Thrombocytes below lower limit of normal or liver enzymes (ALT, AST, GGT, AP) above upper limit of normal at the screening examination
* Subjects with CYP 2C19 PM status

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an open-label, mono-center clinical trial in healthy male subjects applied a two-period, two-treatment, fixed sequence design. Each subject participated in the two trial periods (Visit 2 [Days 1 and 2] and Visit 3 [Days -7 to 2] and received the two treatments in the same sequence in Period 1 the Reference treatment (R) and afterwards in Period 2 the Test treatment (T).
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended one specialist site which would then ensure that they (the subjects) met all inclusion/exclusion criteria. The subjects were not included into the trial if any one of the specific entry criteria were violated.
Period: Period 1 (R)
Arm/Group | BI 409306 (R), Then BI 409306 After Pretreatment With Rifampicin (T)
Started | 15
Completed | 15
Not Completed | 0
Period: Period 2 (T)
Arm/Group | BI 409306 (R), Then BI 409306 After Pretreatment With Rifampicin (T)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set includes all subjects who were entered and dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | BI 409306 (R), Then BI 409306 After Pretreatment With Rifampicin (T)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) is reported.
Time Frame: Within 3 hours (h) before and 0.333h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 11h, 12h, 24h after drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): all subjects in the TS who provided at least one primary or secondary PK parameter not flagged for exclusion due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Least Squares Mean (Standard Error); unit: nanomole*hour/liter (nmol·h/L)
Groups:
- T: BI 409306 + Rifampicin Pretreatment: On Days -7 to -1 / Visit 3 of Period 2 participants were administered rifampicin 600 milligrams (mg) Eremfat® film-coated tablet orally with 240 milliliter (mL) of water once per day during the evenings. Afterwards on Day 1/Visit 3, participants were administered a single dose of 50 mg BI 409306 orally approximately 14 hours after the last rifampicin dose (test treatment, T).
- R: BI 409306: Subjects were administered during Period 1 on Day 1/Visit 2 a single dose of 50 milligrams (mg) of BI 409306 film-coated tablet orally with 240 millilitre (mL) of water (reference treatment, R).
Arm/Group | T: BI 409306 + Rifampicin Pretreatment | R: BI 409306
Number analyzed (Participants) | 15 | 15
nanomole*hour/liter (nmol·h/L) | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 79.05 Standard error is actually geometric standard error. Geometric standard error =1.263. | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 1013.34 Standard error is actually geometric standard error. Geometric standard error =1.263.
Statistical Analysis 1: Comparison: T: BI 409306 + Rifampicin Pretreatment vs R: BI 409306; The main focus is on estimation, therefore no hypothesis was tested. The statistical analysis model for the primary endpoints is an ANOVA (analysis of variance). This model included effects accounting for the following sources of variation: 'subjects' and 'treatment'. The effect 'subjects' will be considered as random, whereas the treatment effect will be considered as fixed. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model; Test type: Other; Geometric mean (gMean) ratio (%) = 7.80, 90% CI 2-sided [5.740 to 10.601], Standard Error of Mean 1.190 — gMean ratio = BI 409306 + Rifampicin pretreatment (T) / BI 409306 (R). Standard Error of the mean is actually the Geometric Standard Error

2. Primary Outcome: Maximum Measured Concentration of BI 409306 in Plasma (Cmax)
Description: Maximum measured concentration of BI 409306 in plasma (Cmax) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nanomole/liter (nmol/L)
Arm/Group | T: BI 409306 + Rifampicin Pretreatment | R: BI 409306
Number analyzed (Participants) | 15 | 15
nanomole/liter (nmol/L) | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 64.49 Standard error is actually geometric standard error. Geometric standard error =1.258 | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 660.29 Standard error is actually geometric standard error. Geometric standard error =1.258
Statistical Analysis 1: Comparison: T: BI 409306 + Rifampicin Pretreatment vs R: BI 409306; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric mean (gMean) ratio (%) = 9.77, 90% CI 2-sided [6.767 to 14.098], Standard Error of Mean 1.232 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 409306 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 409306 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nanomole*hour/liter (nmol·h/L)
Arm/Group | T: BI 409306 + Rifampicin Pretreatment | R: BI 409306
Number analyzed (Participants) | 15 | 15
nanomole*hour/liter (nmol·h/L) | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 83.96 Standard error is actually geometric standard error. Geometric standard error =1.258 | NA (NA) — Least squares mean is actually adjusted geometric mean (gMean). Adjusted geometric mean (gMean)= 1020.71 Standard error is actually geometric standard error. Geometric standard error =1.258
Statistical Analysis 1: Comparison: T: BI 409306 + Rifampicin Pretreatment vs R: BI 409306; Since the main focus is on estimation and not testing, therefore no hypothesis was tested.The statistical analysis model is an ANOVA (analysis of variance) model on the logarithmic scale. This model included effects accounting for the following sources of variation: 'subjects' and 'treatment'. The effect 'subjects' will be considered as random, whereas the treatment effect will be considered as fixed. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model; Test type: Other; Geometric mean (gMean) ratio (%) = 8.23, 90% CI 2-sided [6.081 to 11.126], Standard Error of Mean 1.187 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration through the Residual effect period (REP) until end of trial; up to 14 days
Description: The Adverse Event assessment was reported for Period 1: BI 409306, and for Period 2 separately: rifampicin pretreatment and; BI 409306 subsequent to rifampicin pretreatment.
Groups:
- Test Treatment, T: Rifampicin Pretreatment: On Days -7 to -1 / Visit 3 of Period 2 participants were administered rifampicin 600 mg Eremfat® film-coated tablet orally with 240 mL of water once per day during the evenings (First 7 Days of Period 2).
- Test Treatment, T: BI 409306 Subsequent to Rifampicin Pretreatment: On Days -7 to -1 / Visit 3 of Period 2 participants were administered rifampicin 600 mg Eremfat® film-coated tablet orally with 240 mL of water once per day during the evenings. After on Day 1/Visit 3, participants received a single dose of 50 mg BI 409306 orally approximately 14 hours after the last rifampicin dose (test treatment, T).
Arm/Group | R: BI 409306 | Test Treatment, T: Rifampicin Pretreatment | Test Treatment, T: BI 409306 Subsequent to Rifampicin Pretreatment
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 15/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R: BI 409306 (N=15) | Test Treatment, T: Rifampicin Pretreatment (N=15) | Test Treatment, T: BI 409306 Subsequent to Rifampicin Pretreatment (N=15)
Photopsia (Eye disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 15 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT03151499/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT03151499/SAP_001.pdf